CLINICAL TRIAL: NCT01657097
Title: Allergic Inflammation in Rhinitis Patients Following Nasal Allergen Challenge. Impact on Bronchial Hyperresponsiveness and the Effect of Intranasal Corticosteroid Treatment
Brief Title: Allergic Inflammation in Rhinitis Patients Following Nasal Allergen Challenge
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RHINO97
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- INCS (Experimental): Fluticasone propionate 400 microgram daily
  Interventions: Drug: INCS
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCS
  Arms: INCS
Drug: Placebo
  Arms: Placebo

SUMMARY:
Allergic rhinitis is a common condition caused by inflammation of nasal mucosa. The study was performed to gain information on this inflammation, including effect of intranasal corticosteroid treatment hereupon and potential influence on the lower airways, ie asthma.

The study was randomised, placebo-controlled double-blind in patients, monoallergic to grasspollen, presenting symptoms of rhinitis and asthma during season.

Treatment,ie intranasal corticosteroid or placebo, were given four weeks. After two weeks of treatment intranasal allergen challenge was performed. Measurements were performed during the full study period.

The study was performed out of pollen season.

ELIGIBILITY:
Inclusion Criteria:

* monoallergy to grass
* symptoms of allergic rhinitis for at least the two most recent grasspollen seasons
* asthma symptoms of asthma for at least two of the four most recent grasspollen seasons
* age 18 or older

Exclusion Criteria:

* pregnancy or lactation
* fertile women, not sterilised or using sufficient anticonception
* Corticosteroid treatment (parenteral, oral, inhaled or intranasal) within two months prior to enrolment
* Any other disease, condition or treatment, which to the discretion of the investigator has the potential to interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1997-02; Primary Completion 1997-04 (Actual); Study Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Serum Eosinophil Cationic Protein (ECP) | 1 month

SECONDARY OUTCOMES:
Serum Eosinophil Peroxidase (EPO) | 1 month
Nasal lavage Eosinophil Cationic Protein (ECP) | 1 month
Nasal lavage Eosinophil Peroxidase (EPO) | 1 month
Blood Eosinophils | 1 month

OTHER OUTCOMES:
Bronchial metacholine challenge | 1 month
Acoustic rhinometry | 1 month
Spirometry (Forced Expiratory Volume 1 second (FEV-1)) | 1 month
Nasal symptom score | 1 month
Asthma symptom score | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, MD, Principal Investigator — Department of Respiratory Diseases, Aarhus University Hospital
Locations (1):
- Department of Respiratory Diseases, Aarhus University Hospital, Aarhus, Denmark